CLINICAL TRIAL: NCT06654726
Title: A Phase 2b/3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of Aldafermin in Subjects With Primary Sclerosing Cholangitis (ALPINE-PSC).
Brief Title: A Multi-center Evaluation of Aldafermin in a Randomized, Double-blind, Placebo-controlled Study in Subjects With Primary Sclerosing Cholangitis.
Acronym: ALPINE-PSC
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated by the Sponsor because the FDA advised a trial design change which made it infeasible to continue the study.
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 282-PS-231
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- aldafermin (Experimental): Aldafermin 3mg given subcutaneously, daily, for up to 6 years
  Interventions: Drug: aldafermin
- placebo (Placebo Comparator): Placebo given subcutaneously, daily, for up to 6 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: aldafermin — aldafermin
  Arms: aldafermin
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
A multi-center evaluation of aldafermin in a randomized, double-blind, placebo-controlled study in subjects with Primary Sclerosing Cholangitis.

DETAILED DESCRIPTION:
Evaluation of Efficacy, Safety and Tolerability of Aldafermin in a Phase 2b/3, Randomized, Double-blind, Placebo-controlled, Multi-center Study in Subjects with Primary Sclerosing Cholangitis (ALPINE-PSC)

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give informed consent
2. Confirmed diagnosis of PSC based on either:

   1. Abnormal cholangiography consistent with PSC as measured by MRCP with contrast
   2. Liver biopsy consistent with PSC
3. LSM by VCTE, indicative of at least F2 liver fibrosis stage
4. Laboratory parameters:

   1. TBL ≤2.5 mg/dL unless known for Gilbert's Syndrome
   2. ALT and ALT <5x ULN
   3. MELD score ≤12

Exclusion Criteria:

1. Clinically significant acute or chronic liver disease of an etiology other than PSC
2. Alternate causes of sclerosing cholangitis including IgG4 related sclerosing cholangitis
3. Subjects with moderate to severe hepatic impairment
4. Subjects with moderate to severe renal impairment
5. Placement of bile duct stent or percutaneous bile duct drain within 12 weeks of Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Enhanced Liver Fibrosis Score at Week 96 | 96 Weeks
  Enhanced Liver Fibrosis (ELF) score is a non-invasive blood test derived from the measurement of hyaluronic acid (HA), amino terminal propeptide of type III procollagen (PIIINP), and tissue inhibitor of metalloprotease 1 (TIMP1) using a proprietary algorithm (Siemens). ELF score is a laboratory test, is unitless, and is used as a continuous variable. The minimal ELF score is zero, the maximal ELF score is unknown. The higher the ELF score, the worse the disease outcome.
  ELF is a score on a scale of severity assessment against biopsy-proven fibrosis. A score of <7.7 is none to mild, > 7.7-9.8 is moderate, > 9.8 is severe.